CLINICAL TRIAL: NCT05526612
Title: The Effects of Motor Imagery Training and Physical Practice on Upper Extremity Motor Function in Patients With Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Nisa Nur SOYSAL, Principal Investigator,Physical Therapist, Biruni University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B-SOYSAL-001
Record Dates: First submitted 2022-08-31; First posted 2022-09-02 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Stroke
Keywords: Stroke; Motor imagery; Physical practice; Bobath therapeutic approach
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Parallel Assignment (Outcomes Assessor)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Motor imagery and Bobath Therapeutic Approach (BTA+MI)
  Interventions: Other: Group 1 Motor imagery and Bobath Therapeutic Approach (BTA+MI)
- Group 2 (Experimental): Motor imagery, Bobath Therapeutic Approach and Physical practice (BTA+MI+PP)
  Interventions: Other: Group 2 Motor imagery, Bobath Therapeutic Approach and Physical practice (BTA+MI+PP)

INTERVENTIONS:
Other: Group 1 Motor imagery and Bobath Therapeutic Approach (BTA+MI) — Motor imagery (MI) is the mental rehearsal of motor abilities to improve function. Without revealing any movement in the body, the representation of the movement is created in the mind, the person imagines that he/she is performing the movement. Eating activity will be applied in motor imagery. Individualized therapy sessions in the Bobath Therapeutic Approach will also be received by the Physiotherapist along with Motor imagery. 2 days a week, 30 minutes session will be applied for a total of 8 weeks.
  Arms: Group 1
Other: Group 2 Motor imagery, Bobath Therapeutic Approach and Physical practice (BTA+MI+PP) — Individualized therapy sessions in the Bobath Therapeutic Approach with motor imagery will be performed by the physiotherapist, and in addition to these, 5 repetitions of the eating activity used in motor imagery will be practiced. 2 days a week, 30 minutes session will be applied for a total of 8 weeks.
  Arms: Group 2

SUMMARY:
The aim of the study is to compare the effects of specific functional task-oriented motor imagery training combined with the Bobath Therapeutic Approach and physical practice after imagery on upper extremity motor function in stroke patients.

DETAILED DESCRIPTION:
Motor imagery (MI) is the mental rehearsal of motor abilities to improve function. Thus, imagery provides both the learning of the new movement and the improvement of the quality of movement by repeating the known activities.the investigators These neurophysiological findings obtained in recent years have popularized the use of motor imagery approach in the rehabilitation of stroke patients.

32 stroke patients aged 50-75 years will be included in the study. Cases will be randomized into 2 groups.

In our study, a treatment program will be applied with a physiotherapist for a total of 8 weeks, 2 days a week. The first group in the treatment program; Motor imagery will be performed with the Bobath Therapeutic Approach (BTA+MI) and the second group will be physical practice of imagery activities after motor imagery with the Bobath Therapeutic Approach (BTA+MI+PP). Motor imagery activity was determined as 'eating activity'.

The desired goal as a result of our work; the investigators think that motor imagery training on eating activity of stroke patients and physical practice used together will improve both the achievement of eating activity and upper extremity motor function.

ELIGIBILITY:
Inclusion Criteria:

* A maximum of 24 months have passed since the stroke,
* Unilateral involvement,
* Getting a score of 21 and above in the Mini Mental Test,
* Getting a score of 22 and above in the Fugl-Meyer Test,
* Ability to understand and follow simple verbal commands,
* Stage 4 or 5 according to Brunnstrom Upper Extremity Stages,
* Spasticity 1 or 1+ according to the Modified Ashworth Scale,
* Having signed the Informed Consent Form.

Exclusion Criteria:

* Patients with visual and hearing impairments that would interfere with work.
* Having pain and limitation of joint movement that may prevent performing the given tasks.
* Having any neurological disorder other than stroke.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-07-13 (Actual); Primary Completion 2022-08-13 (Actual); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
The Fugl-Meyer Upper Extremity Scale (FMUE) | The first assessment was evaluated at baseline and the second assessment evaluated change after 8 weeks of rehabilitation
  Fugl-Meyer upper extremity (FMUE) Scale scores is an index to assess the sensorimotor impairment in individuals who had stroke.
  The motor section score ranges from 0 to 66, and the score related to exteroceptive and proprioceptive sensitivity ranges from 0 to 12. The lowest and highest scores correspond to worse and better function.
Time in minutes to perform a motor task | The first assessment was evaluated at baseline and the second assessment evaluated change after 8 weeks of rehabilitation
  The video will be recorded while the patient is performing the eating activity.
The Motor Activity Log-28 (MAL-28) | The first assessment was evaluated at baseline and the second assessment evaluated change after 8 weeks of rehabilitation
  Motor Activity Log is developed to determine the frequency and quality of use of the affected arm It consists of two scales that question how often the affected side's upper extremity is used for each activity during the 28-day activity (Usage Quantity Scale) and how well it can perform the activity if it uses it. On both scales, the patient scores between 0-5. The score that can be obtained is between 0-5 points and the high score indicates good frequency of use and good quality of movement.
Wolf Motor Function Test (WMFT) | The first assessment was evaluated at baseline and the second assessment evaluated change after 8 weeks of rehabilitation
  The Wolf Motor Function Test (WMFT) quantifies upper extremity (UE) motor ability through timed and functional tasks. When administering the WMFT, the examiner should test the less-affected UE followed by the most affected side. Items should be performed as quickly as possible; a maximum of 120 second per task is allowed . The first 6 items involve timed functional tasks, items 7-14 are measures of strength, and the remaining 9 items consist of analyzing movement quality when completing various tasks.

SECONDARY OUTCOMES:
Demographic Characteristic of Participants | 1 week before the first treatment session
  The general demographic information of participants such as gender, age, body mass index will be recorded in a form created by investigators.
Assessment of Quality of Life | The first assessment was evaluated at baseline and the second assessment evaluated change after 8 weeks of rehabilitation
  Nottingham Extended Activities of Daily Living (NEADL)
  It is a simple, self-administered questionnaire that can be completed by the patient in approximately 10 min; it provides an extended ADL score that is highly correlated with more complex, self-reported interviewer-administered measures of disability.
The Brunnstrom Stages | Baseline
  The brunnstrom stages is one of the most well-known stroke recovery stages which is also known as the Brunnstrom approach. The motor recovery of hemiplegia was classified by Brunnstrom in 6 stages.
Spasticity Evaluation | Baseline
  Modified Ashworth Scale (MAS)
  It is used to measure spasticity which ranges from 0-4.
The Kinesthetic and Visual Imagery Questionnaire (KVIQ) | The first assessment was evaluated at baseline and the second assessment evaluated change after 8 weeks of rehabilitation
  The KVIQ assesses on a five-point ordinal scale the clarity of the image (visual: V subscale) and the intensity of the sensations (kinesthetic: K subscale) that the subjects are able to imagine from the first-person perspective.

CONTACTS AND LOCATIONS:
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-09-02): https://cdn.clinicaltrials.gov/large-docs/12/NCT05526612/Prot_SAP_ICF_000.pdf